CLINICAL TRIAL: NCT04895410
Title: A Phase 1b, Dose Escalation and Expansion Study of Lemzoparlimab With or Without Dexamethasone and in Combination With Anti-Myeloma Regimens for the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study to Assess Adverse Events and Change in Disease Activity of Intravenous (IV) Lemzoparlimab With or Without Oral/IV Dexamethasone and in Combination With Oral/IV/Subcutaneous Anti-Myeloma Regimens in Adult Participants With Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-917; 2021-001067-24 (EudraCT Number)
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
Keywords: Lemzoparlimab; ABBV-IMAB-TJC4; Relapsed or refractory multiple myeloma (R/R MM); Cancer; TJ011133; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Neoplasms | interventions — Dexamethasone; carfilzomib; pomalidomide; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Dose Escalation: Lemzoparlimab (Experimental): Participants will receive lemzoparlimab in 28 day cycles.
  Interventions: Biological: Lemzoparlimab
- Dose Escalation: Lemzoparlimab + Pomalidomide + Dexamethasone (Experimental): Participants will receive lemzoparlimab + pomalidomide + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Drug: Pomalidomide
- Dose Escalation: Lemzoparlimab + Carfilzomib + Dexamethasone (Experimental): Participants will receive lemzoparlimab + carfilzomib + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Drug: Carfilzomib
- Dose Escalation: Lemzoparlimab + Daratumumab + Dexamethasone (Experimental): Participants will receive lemzoparlimab + daratumumab + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Biological: Daratumumab
- Dose Expansion: Lemzoparlimab (Experimental): Participants will receive lemzoparlimab at recommended dose determined in Dose Escalation portion in 28 day cycles.
  Interventions: Biological: Lemzoparlimab
- Dose Expansion: Lemzoparlimab + Dexamethasone (Experimental): Participants will receive lemzoparlimab at recommended dose determined in Dose Escalation portion + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone
- Dose Expansion: Lemzoparlimab + Pomalidomide + Dexamethasone (Experimental): Participants will receive lemzoparlimab at recommended dose determined in Dose Escalation portion + pomalidomide + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Drug: Pomalidomide
- Dose Expansion: Lemzoparlimab + Carfilzomib + Dexamethasone (Experimental): Participants will receive lemzoparlimab at recommended dose determined in Dose Escalation portion + carfilzomib + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Drug: Carfilzomib
- Dose Expansion: Lemzoparlimab + Daratamumab + Dexamethasone (Experimental): Participants will receive lemzoparlimab at recommended dose determined in Dose Escalation portion + daratamumab + dexamethasone in 28 day cycles.
  Interventions: Biological: Lemzoparlimab; Drug: Dexamethasone; Biological: Daratumumab

INTERVENTIONS:
Biological: Lemzoparlimab — Intravenous (IV) infusion
  Other Names: TJ011133
Drug: Dexamethasone — Oral tablet or IV infusion/injection
  Arms: Dose Escalation: Lemzoparlimab + Carfilzomib + Dexamethasone; Dose Escalation: Lemzoparlimab + Daratumumab + Dexamethasone; Dose Escalation: Lemzoparlimab + Pomalidomide + Dexamethasone; Dose Expansion: Lemzoparlimab + Carfilzomib + Dexamethasone; Dose Expansion: Lemzoparlimab + Daratamumab + Dexamethasone; Dose Expansion: Lemzoparlimab + Dexamethasone; Dose Expansion: Lemzoparlimab + Pomalidomide + Dexamethasone
Drug: Carfilzomib — IV infusion
  Arms: Dose Escalation: Lemzoparlimab + Carfilzomib + Dexamethasone; Dose Expansion: Lemzoparlimab + Carfilzomib + Dexamethasone
Drug: Pomalidomide — Oral capsule
  Arms: Dose Escalation: Lemzoparlimab + Pomalidomide + Dexamethasone; Dose Expansion: Lemzoparlimab + Pomalidomide + Dexamethasone
Biological: Daratumumab — Subcutaneous (SC) injection
  Arms: Dose Escalation: Lemzoparlimab + Daratumumab + Dexamethasone; Dose Expansion: Lemzoparlimab + Daratamumab + Dexamethasone

SUMMARY:
Multiple myeloma (MM) accounts for more than 10% of all blood cancers and 1% of all cancers. The purpose of this study is to assess how safe lemzoparlimab is and how lemzoparlimab moves through the body of adult participants with MM when given with or without dexamethasone, and in combination with other anti-myeloma regimens. Adverse events and change in disease activity will be assessed.

Lemzoparlimab is an investigational drug being developed for the treatment of relapsed/refractory (R/R) MM. Study doctors put the participants in groups called treatment arms. Two different dose levels of lemzoparlimab will be explored. Each treatment arm receives a different treatment combination depending on stage of the study and eligibility. This study will include a dose escalation phase to determine the best dose of lemzoparlimab, followed by a dose expansion phase to confirm the dose. Approximately 163 adult participants with R/R MM will be enrolled in the study in approximately 60 sites worldwide.

In the Dose Escalation arms, participants will receive intravenous (IV) lemzoparlimab with or without dexamethasone (oral/IV) in combination with pomalidomide (oral) or carfilzomib (IV) or subcutaneous (SC) daratumumab in 28-day cycles. In the Dose Expansion arms, participants will receive lemzoparlimab (IV) alone or with dexamethasone (oral/IV) in combination with pomalidomide (oral) or carfilzomib (IV) or daratumumab (SC) in 28-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed/refractory (R/R) multiple myeloma (MM) with documented evidence of progression during or after the participant's last treatment regimen based on the investigator's determination of the International Myeloma Working Group (IMWG) criteria.

  * Relapsed defined as previously treated myeloma that progresses and requires initiation of salvage therapy, but does not meet criteria for refractory myeloma.
  * Refractory defined as disease that is nonresponsive (failure to achieve minimal response or development of progressive disease) while on primary or salvage therapy, or progresses within 60 days of last therapy.
* Measurable disease per the protocol within 28 days prior to enrollment.
* Arm A - Lemzoparlimab with or without Dexamethasone

  * For Both Escalation and Expansion Phase, participant must have refractory to 3 prior lines of treatment of anti-myeloma treatments, as outlined in the protocol.
* Arm B - Lemzoparlimab + Pomalidomide-Dexamethasone

  * For Escalation Phase - Participant must have received at least 3 prior lines of therapy, as outlined in the protocol.
  * For Expansion Phase- Participant must have received at least 2 prior line of therapy, as outlined in the protocol.
* Arm C - Lemzoparlimab + Carfilzomib-Dexamethasone

  * For Escalation Phase- Participant must have received at least 3 prior lines of therapy as outlined in the protocol.
  * For Expansion Phase- Participant must have received at least 1 prior line of therapy.
* Arm D - Lemzoparlimab + Daratumumab-Dexamethasone -- For Both Escalation and Expansion Phase - Participant must: --- Have received at least 3 prior lines of therapy, as outlined in the protocol.

Exclusion Criteria:

* Arm B - Lemzoparlimab + Pomalidomide-Dexamethasone

  * For Both Escalation and Expansion Phase participant must have had no prior treatment with pomalidomide.
* Arm C - Lemzoparlimab + Carfilzomib-Dexamethasone

  * For Both Escalation and Expansion Phase - prior treatment with carfilzomib.
* Arm D - Lemzoparlimab + Daratumumab-Dexamethasone

  * For Both Escalation and Expansion Phase - prior treatment with daratumumab or other anti-CD38 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) of Lemzoparlimab With or Without Dexamethasone and in Combination With Anti-myeloma Regimens in Participants With Relapsed/Refractory (R/R) Multiple Myeloma (MM) | Up to 28 days after study drug administration
  DLT events as described in the protocol will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Best Overall Response of Documented Partial Response (PR) or Better | Up to approximately 2 years
  Best overall response is defined as achieving documented PR or better at two consecutive disease assessments during the study, according to International Myeloma Working Group (IMWG) 2016 criteria.
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the first dose of study drug to the first documented progressive disease (PD) or death due to any cause, whichever occurs first.
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from first documented response (PR or better) to the first documented PD or death due to MM, whichever occurs first.
Time to Progression (TTP) | Up to approximately 2 years
  TTP is defined as the time from the first dose of study drug to the first documented PD or death due to MM, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- United States (12):
  - Sylvester Comprehensive Cancer Center /ID# 228817, Miami, Florida
  - Moffitt Cancer Center /ID# 229939, Tampa, Florida
  - Norton Cancer Institute - St Matthews /ID# 229319, Louisville, Kentucky
  - Tulane Cancer Center Clinic /ID# 229832, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 229309, Ann Arbor, Michigan
  - Henry Ford Health System /ID# 230341, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey /ID# 230174, New Brunswick, New Jersey
  - Columbia University Medical Center /ID# 229971, New York, New York
  - Duke University Hospital /ID# 229564, Durham, North Carolina
  - Wake Forest Baptist Health /ID# 229996, Winston-Salem, North Carolina
  - Perelman Center for Advanced Medicine - /ID# 228693, Philadelphia, Pennsylvania
  - University of Virginia /ID# 229396, Charlottesville, Virginia
- Australia (2):
  - The Queen Elizabeth Hospital /ID# 229345, Woodville South, South Australia
  - Alfred Health /ID# 229347, Melbourne, Victoria
- France (4):
  - HCL - Hôpital Lyon Sud /ID# 229834, Pierre-Bénite, Auvergne-Rhône-Alpes
  - CHU de Nantes, Hotel Dieu -HME /ID# 228559, Nantes, Pays de la Loire Region
  - CHU Poitiers - La milétrie /ID# 229833, Poitiers, Poitou-Charentes
  - Hopital Henri Mondor /ID# 228562, Créteil
- Asklepios Klinik Altona /ID# 229143, Hamburg, Germany
- Israel (6):
  - The Chaim Sheba Medical Center /ID# 229483, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 229478, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 229485, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 229477, Jerusalem
  - Meir Medical Center /ID# 229480, Kfar Saba
  - Rabin Medical Center /ID# 229488, Petah Tikva
- University Hospital Kyoto Prefectural University of Medicine /ID# 241833, Kyoto, Kyoto, Japan
- Spain (6):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 229356, Santiago de Compostela, A Coruna
  - Hospital Unversitario Marques de Valdecilla /ID# 229354, Santander, Cantabria
  - Hospital Parc de Salut del Mar /ID# 229371, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 229369, Barcelona
  - Hospital Universitario Reina Sofia /ID# 229388, Córdoba
  - Hospital Universitario 12 de Octubre /ID# 229355, Madrid

IPD SHARING:
Plan to Share IPD: No